CLINICAL TRIAL: NCT06271824
Title: Developing and Piloting a Tailored Self-Compassion Program to Enhance the Well-Being of Informal Caregivers of Children With Physical Disabilities
Brief Title: Self-Compassion to Enhance the Well-Being of Caregivers of Children With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-1519
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-03

CONDITIONS: Stress; Caregiver Burden; Anxiety; Depressive Symptoms
MeSH Terms: conditions — Caregiver Burden; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Live, online socio-emotional group course
  Interventions: Behavioral: Self-Compassion Based Resilient Caregiving Course

INTERVENTIONS:
Behavioral: Self-Compassion Based Resilient Caregiving Course — The Resilience Habits for Caregivers Course is a live, online, weekly 6 session program lasting 1.5 hours per session. The structure contains didactics, group discussions, guided exercises, and practices facilitated by a certified self-compassion instructor. Topics covered include: (1) noticing and accepting emotions (including conflicting emotions); (2) cultivating curiosity and self-compassion; (3) relating skillfully to difficult thoughts; (4) savoring and gratitude practices.

SUMMARY:
The goal of this clinical trial is to test the feasibility, acceptability and preliminary social/emotional well-being outcomes of a tailored, online self-compassion-based resilience course for caregivers of children with physical disabilities. The main questions it aims to answer are:

1. Is the online resilience course feasible and acceptable to caregivers of children with physical disabilities?
2. Is participation in the resilience course associated with improvements in caregiver stress, anxiety, depression, burden, caregiver uplifts, self-compassion, emotion regulation and/or resilience?

Participants will complete a screening, a verbal consent process and an electronic pre-course survey. Then, they will participate in a 6-session weekly online course with other caregivers and led by a certified Mindful Self-Compassion instructor. The course has been created with feedback from caregivers and includes skills for recognizing and coping with difficult emotions while connecting with others who have similar caregiving experiences. After the course, participants will repeat the electronic survey and will provide feedback on the course during a live, online feedback session.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is at least 18 years old
* Caregiver reads and speaks in English
* Caregiver is a primary caregiver to a child aged 2-17 with a moderate to severe chronic physical disability (child requires assistance or adapted methods for mobility (e.g., walking, transfers) and at least 1 other functional area (e.g., toileting, feeding, communication))

Exclusion Criteria:

* Caregiver has no access to the internet/Zoom
* Caregiver has been hospitalized in the last year for mental health treatment
* Caregiver has a history of psychosis (e.g., schizophrenia)
* Caregiver will miss 2 or more class sessions due to scheduling conflicts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who withdraw from course | Across 6 weeks of intervention
  The study records will indicate withdrawal status (Yes or No) for each enrolled participant who has attended at least 1 intervention session; Calculated by: number who withdraw/total number enrolled X 100
Percentage of participants who attend at least 4 of 6 intervention sessions | Across 6 weeks of intervention
  The study records will indicate weekly attendance at each session (Yes or No) for each enrolled participant who has attended at least 1 intervention session. Calculated by: number who attend at least 4 of 6 sessions/total number enrolled X 100
Percentage of participants who rate the course as "acceptable" or "completely acceptable" | 6 weeks
  The Theoretical Framework of Acceptability includes 7-items regarding intervention acceptability on a scale of 1 to 5, scores range 7-35, higher numbers indicate greater acceptability. This general acceptability item will be used to assess overall acceptability of the course. Calculated by: number of participants who endorse "acceptable" or "completely acceptable"/total number of respondents X 100
Percentage of intervention topics covered | Across 6 weeks of intervention
  A research assistant in attendance will use a fidelity checklist to assess if intended topics are covered each session (Yes/No). Calculated by number of topics covered/total number of topics intended to be covered X 100

SECONDARY OUTCOMES:
Mean Change in Perceived Stress as Measured by the Perceived Stress Scale (PSS-10 item) at 6 weeks | Baseline and 6 weeks
  The PSS is a validated 10 item scale assessing the degree to which situations in one's life are perceived as stressful assessed over the last 7 days; scale ranges from 0=never to 4=very often; total scores range from 0 to 40 with higher scores indicating higher stress.
Mean Change in Resilience as measured by the Connor-Davidson Resilience Scale-10 at 6 weeks | Baseline and 6 weeks
  The Connor-Davidson Resilience Scale is an 10-item measure of resilience and hardiness. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4, total scores range from 0 to 40, and higher scores indicate higher resilience.
Mean Change in Anxiety as measured by the PROMIS-SF 7-item Anxiety Scale at 6 weeks | Baseline and 6 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1. 0 - Anxiety 7a questionnaire includes 7 questions related to anxious mood in the past 7 days. Each question is rated on a five-point scale from 1=Never to 5=Always, with total scores ranging from 7-35 and higher scores indicating higher anxiety levels.
Mean Change in Depressive symptoms as measured by the PROMIS-SF 8-item Depression Scale at 6 weeks | Baseline and 6 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Depression scale measures depressive symptoms in the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Mean Change in Self-Compassion as measured by the Self-Compassion Scale-Short form (SCS-SF) at 6 weeks | Baseline and 6 weeks
  The SCS-SF is a 12 item scale that measures how often one is self-compassionate. Each item is rated on a 5-point scale from 1=almost never to 5=almost always with a range in score from 8 to 40 with higher scores indicating greater frequency of self-compassion.
Mean Change in Caregiver Burden as measured by the 12-item Zarit Caregiver Burden Scale (ZBI-12) at 6 weeks | Baseline and 6 weeks
  The ZBI-12 is a 12 item scale measuring caregiver burden. Each item is rated from 0 (never) to 4 (nearly always) with a range from 0 to 48 and higher scores indicating higher burden.
Mean Change in Caregiver Uplifts as measured by the Uplifts subscale of the Revised Burden Measure at 6 weeks | Baseline and 6 weeks
  The Uplifts subscale measures positive aspects of caregiving using 6 items answered in a 5-point response scale ranging from 1 (Not at all) to 5 (A great deal). Scores range from 6-30, with higher scores indicating higher degrees of positive experiences in caregiving.
Mean Change in Difficulties with Emotion Regulation as measured by the Difficulties in Emotion Regulation-Short Form Scale | Baseline and 6 weeks
  The Difficulties in Emotion Regulation scale measures difficulties with regulation of emotions using 18-items representing 6 subscales (strategies, nonacceptance, impulse, goals, awareness and clarity) answered in a 5-point response scale ranging from 1 (Almost never) to 5 (almost always). Total scores range from 18- 90 with higher scores indicating higher levels of difficulty with emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lathren, MD, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No